CLINICAL TRIAL: NCT04344665
Title: Post Discharge After Surgery Virtual Care With Remote Automated Monitoring Technology (PVC-RAM) Trial
Acronym: PVC-RAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: v5.0, 2020.09.12
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Perioperative Complication; COVID
Keywords: Virtual care; Remote monitoring; Days alive at home

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Care and Remote Automated Monitoring (Experimental)
  Interventions: Other: Virtual Care and Remote Automated Monitoring
- Standard Care (No Intervention)

INTERVENTIONS:
Other: Virtual Care and Remote Automated Monitoring — Patients will measure daily vitals (blood pressure, heart rate, respiratory rate, oxygen saturation, temperature, weight) with remote monitoring technology and complete recovery surveys daily in home after discharge from hospital. Patients will interact with a virtual nurse daily on days 1-15 and every other day from days 16-30. If the patient's RAM measurements exceed predetermined thresholds, the patient reports specific symptoms (e.g., shortness of breath), a drug error is identified, or the virtual nurse has concerns about the patient's health that they cannot resolve, the virtual nurse will escalate care to a pre-assigned and available physician. Physicians will add or modify treatments as needed, and if required, they will have the patient come to an outpatient facility for evaluation or management. Via secure video or text messaging, patients will also have access to a virtual nurse at night, for any urgent issues.
  Arms: Virtual Care and Remote Automated Monitoring

SUMMARY:
The Post discharge after surgery Virtual Care with Remote Automated Monitoring technology (PVC-RAM) Trial is a multicentre, parallel group, superiority, randomized controlled trial to determine the effect of virtual care with remote automated monitoring (RAM) technology compared to standard care on days alive at home during the 30-day follow-up after randomization, in adults who have undergone semi-urgent (e.g., oncology), urgent (e.g., hip fracture), or emergency (e.g., ruptured abdominal aortic aneurysm) surgery. It will also determine, during the first 30 days, the effect of virtual care with RAM technology on several secondary outcomes, including: 1. hospital re-admission; 2. emergency department visit; 3. urgent-care centre visit; 4. acute-hospital care (i.e., a composite of hospital re-admission and emergency department or urgent-care centre visit) 5. brief acute-hospital care (i.e., acute-hospital care that lasts <24 hours); 6. all-cause hospital days; 7. medication error detection; 8. medication error correction; and 9. death. An additional secondary objective is to determine the effect of virtual care with RAM technology on pain at 7, 15, and 30 days and 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥40 years of age;
2. have undergone same-day or inpatient semi-urgent, urgent, or emergency surgery and are being discharged home or are within 24 hours after discharge home, as long as they have not had acute-hospital care since their discharge; and
3. provide informed consent to participate.

Exclusion Criteria:

1. underwent same-day surgery and the surgeon or anesthesiologist believe the case reflects a traditional same-day surgery case with a low likelihood of needing acute-hospital care;
2. went to rehabilitation or convalescent care for more than 7 days after undergoing surgery;
3. are unable to communicate with research staff, complete study surveys, or undertake an interview using a tablet computer due to a cognitive, language, visual, or hearing impairment; or
4. reside in an area without cellular network coverage and no home Wi-Fi.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Days alive at home | 30 Days (after randomization); 6 months (after randomization)
  Days alive at home are the number of days patients spend at their usual residence - be it a house or apartment, a group home or shelter, a seniors residence, or a nursing home - or at a community residence of a relative, friend, or acquaintance without, during that day, being admitted to a hospital or visiting an emergency department or urgent-care centre. Thus, patients lose days alive at home if 1. patients go to an emergency department or urgent-care centre; 2. they become inpatients at a hospital or rehabilitation or convalescence-care facility; or 3. they die.

SECONDARY OUTCOMES:
Hospital re-admission | 30 Days (after randomization); 6 months (after randomization)
Emergency Department visit | 30 Days (after randomization); 6 months (after randomization)
Urgent Care centre visit | 30 Days (after randomization); 6 months (after randomization)
Brief acute hospital care | 30 Days (after randomization); 6 months (after randomization)
Medication error detection | Days 1, 7, 8, 15, 22 and 30 Days (after randomization in the intervention arm), 30 Days (after randomization in the standard care arm and collected on day 31)
  Medication errors include mistakes in medication prescribing, transcribing, dispensing, administering, or monitoring due to preventable events or actions taken by a patient, caregiver, or healthcare worker. Medication errors include: drug omission (i.e., patient did not take a drug they were supposed to take), drug commission (i.e., patient taking a drug they were not supposed to take), duration error, dosing error, frequency error, route error, and timing error. We will record all drug errors identified and also report whether they resulted in harm.
Medication error correction | Days 1, 7, 8, 15, 22 and 30 Days (after randomization in the intervention arm), 30 Days (after randomization in the standard care arm and collected on day 31)
  Any medication error that is corrected.
Death | 30 Days (after randomization); 6 months (after randomization)
  All cause mortality
Participant Pain | 7 Days (after randomization); 15 Days (after randomization); 30 Days (after randomization); 6 months (after randomization)
  Assessed using the Brief Pain Inventory Short Form (BPI-SF)
Acute hospital care | 30 Days (after randomization); 6 months (after randomization)
  Composite of hospital re-admission and emergency department or urgent-care centre visit
All-cause hospital days | 30 Days (after randomization); 6 months (after randomization)
  If a patient is admitted to the hospital for any reason anytime between midnight and 23:59 on a given day, this will count as a day in hospital.

OTHER OUTCOMES:
Health services utilization-related costs | 30 Days (after randomization); 6 months (after randomization)
  Data on hospital re-admission, healthcare utilization, and costs of health service utilization will be obtained from the Institute for Clinical Evaluative Sciences (ICES) data repository
Patient level cost of recovery | 30 Days (after randomization)
  Assessment performed using the Ambulatory Home Care Record
Re-operation | 30 Days (after randomization); 6 months (after randomization)
  Any surgical procedure undertaken for any reason (e.g., wound dehiscence, infection)
Arrythmia resulting in electrical cardioversion | 30 Days (after randomization); 6 months (after randomization)
  Arrythmia resulting in electrical cardioversion
Acute renal failure resulting in dialysis | 30 Days (after randomization); 6 months (after randomization)
  Acute renal failure resulting in dialysis
Respiratory failure | 30 Days (after randomization); 6 months (after randomization)
  Patient intubated or put on bilevel positive airway pressure (BiPAP).
Infection | 30 Days (after randomization); 6 months (after randomization)
  Infection
Surgical site infection | 30 Days (after randomization); 6 months (after randomization)
Life-threatening bleed | 30 Days (after randomization); 6 months (after randomization)
Major bleed | 30 Days (after randomization); 6 months (after randomization)
Critical organ bleed | 30 Days (after randomization); 6 months (after randomization)
Ileus | 30 Days (after randomization); 6 months (after randomization)
Myocardial Infarction | 30 Days (after randomization); 6 months (after randomization)
Clinically important atrial fibrillation | 30 Days (after randomization); 6 months (after randomization)
Symptomatic proximal venous thrombo-embolism | 30 Days (after randomization); 6 months (after randomization)
Stroke | 30 Days (after randomization); 6 months (after randomization)
Non-fatal cardiac arrest | 30 Days (after randomization); 6 months (after randomization)
Clostridium difficile-associated diarrhea | 30 Days (after randomization); 6 months (after randomization)
Indwelling device | 30 Days (after randomization); 6 months (after randomization)
COVID-19 Infection | 30 Days (after randomization); 6 months (after randomization)
Delirium | 30 Days (after randomization); 6 months (after randomization)
  Positive history of delirium in hospital health records, positive 3D-CAM assessment, or FAM-CAM assessment. Assessments performed by telephone or in person.
Surgeon, family physician, or specialist in-person clinic visit | 30 Days (after randomization); 6 months (after randomization)
Sepsis | 30 Days (after randomization); 6 months (after randomization)
Acute Heart Failure | 30 Days (after randomization); 6 months (after randomization)
Surgeon, family physician, or specialist virtual visit | 30 Days (after randomization); 6 months (after randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGillion, PhD, Principal Investigator — McMaster University, Population Health Research Institute; PJ Devereaux, PhD, Principal Investigator — McMaster University, Population Health Research Institute
Locations (7):
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Hamilton General Hospital, Hamilton
  - Juravinski Hospital, Hamilton
  - St. Joseph's Healthcare Hamilton, Hamilton
  - Kingston Health Sciences Centre, Kingston
  - London Health Sciences Centre, London

IPD SHARING:
Plan to Share IPD: Yes
The Population Health Research Institute (PHRI) is the sponsor of this trial. The PHRI believes the dissemination of clinical research results is vital and sharing of data is important. PHRI prioritises access to data analyses to researchers who have worked on the trial for a significant duration, have played substantial roles, and have participated in raising the funds to conduct the trial. PHRI balances the length of the research study, and the intellectual and financial investments that made it possible with the need to allow wider access to the data collected. Data will be disclosed only upon request and approval of the proposed use of the data by a Review Committee. Data are available to the journal for evaluation of reported analyses. Regarding the ICES data, while data sharing agreements prohibit ICES from making the data set publicly available, access can be granted to those who meet prespecified criteria for confidential access, available at www.ices.on.ca/DAS.

REFERENCES:
- [Derived] McGillion MH, Parlow J, Borges FK, Marcucci M, Jacka M, Adili A, Lalu MM, Ouellette C, Bird M, Ofori S, Roshanov PS, Patel A, Yang H, O'Leary S, Tandon V, Hamilton GM, Mrkobrada M, Conen D, Harvey V, Lounsbury J, Mian R, Bangdiwala SI, Arellano R, Scott T, Guyatt GH, Gao P, Graham M, Nenshi R, Forster AJ, Nagappa M, Levesque K, Marosi K, Chaudhry S, Haider S, Deuchar L, LeBlanc B, McCartney CJL, Schemitsch EH, Vincent J, Pettit SM, DuMerton D, Paulin AD, Simunovic M, Williams DC, Halman S, Harlock J, Meyer RM, Taylor DA, Shanthanna H, Schlachta CM, Parry N, Pichora DR, Yousuf H, Peter E, Lamy A, Petch J, Moloo H, Sehmbi H, Waggott M, Shelley J, Belley-Cote EP, Devereaux PJ; PVC-RAM-1 Investigators. Post-discharge after surgery Virtual Care with Remote Automated Monitoring-1 (PVC-RAM-1) technology versus standard care: randomised controlled trial. BMJ. 2021 Sep 30;374:n2209. doi: 10.1136/bmj.n2209. PMID 34593374
- [Derived] McGillion MH, Parlow J, Borges FK, Marcucci M, Jacka M, Adili A, Lalu MM, Yang H, Patel A, O'Leary S, Tandon V, Hamilton GM, Mrkobrada M, Ouellette C, Bird M, Ofori S, Conen D, Roshanov PS, Harvey V, Guyatt GH, Le Manach Y, Bangdiwala SI, Arellano R, Scott T, Lounsbury J, Taylor DA, Nenshi R, Forster AJ, Nagappa M, Lamy A, Peter E, Levesque K, Marosi K, Chaudhry S, Haider S, Deuchar L, LeBlanc B, McCartney CJL, Schemitsch EH, Vincent J, Pettit SM, Paul J, DuMerton D, Paulin AD, Simunovic M, Williams DC, Halman S, Schlachta CM, Shelley J, Harlock J, Meyer RM, Graham M, Shanthanna H, Parry N, Pichora DR, Yousef H, Moloo H, Sehmbi H, Waggott M, Belley-Cote EP, Whitlock R, Devereaux PJ; PVC-RAM Investigators. Post Discharge after Surgery Virtual Care with Remote Automated Monitoring Technology (PVC-RAM): protocol for a randomized controlled trial. CMAJ Open. 2021 Mar 2;9(1):E142-E148. doi: 10.9778/cmajo.20200176. Print 2021 Jan-Mar. PMID 33653769